CLINICAL TRIAL: NCT02169167
Title: Comparison of Resin Salve and Conventional Octenidine in Patients With Neuropathic Diabetic Foot Ulcers - a Prospective, Randomized and Controlled Clinical Trial
Brief Title: Comparison of Resin Salve and Octenidine in Patients With Neuropathic Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Janne J. Jokinen (Other)
Collaborators: Repolar Pharmaceuticals Oy (Industry)
Responsible Party: Sponsor-Investigator, Janne J. Jokinen, MD, PhD, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NKBBN/75/2014; NKBBN/75/2014 (Other: Gdansk University Hospital)
Record Dates: First submitted 2014-06-19; First posted 2014-06-23 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Diabetes Mellitus; Diabetes Complications; Diabetic Neuropathies; Wound Infection
Keywords: Diabetes complications; Diabetic foot; Foot ulcer; Wound healing; Wound infection
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Complications; Diabetic Neuropathies; Wound Infection; Diabetic Foot; Foot Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resin salve treatment (Experimental): The resin salve may be spread directly onto the diabetic ulcer, after which the area is covered with a bandage suitable for local wound care. The bandage prohibits salve from moving away from the ulcer area. If the skin condition is more widespread or contains cavities or fistulae, the salve may be spread as a film with a thickness of at least 1 mm onto a gauze or gauze ribbon that is then used to fill the cavity or fistulae channel. Bandages are changed every 1-3 days, depending on the degree of infection and amount of ulcer secretion.
  Interventions: Device: Resin salve treatment
- Octenidine treatment (Active Comparator): Octenidine treatment is implemented with the similar manner as resin salve treatment by using sterile gauze that is impregnated with the octenidine dihydrochloride.
  Interventions: Device: Octenidine treatment

INTERVENTIONS:
Device: Resin salve treatment — Resin is collected in the municipality of Kolari, Finland, from the trunks of full-grown Norway spruce (Picea acies) trees. Bark and other impurities are removed mechanically. The resin is then liquefied and purified by filtering. Resin salve is composed of a 10% (w/w) mixture of purified spruce resin in a standardized salve base. None of the components of the salve base have antibacterial properties. Resin salve is produced from the pure resin to the final product in accordance with the Good Manufacturing Standards (GMP) and it holds the European CE mark (Abilar 10% Resin Salve, Repolar Ltd., Espoo, Finland, CE 0537).
  Other Names: Abilar 10% Resin Salve
  Arms: Resin salve treatment
Device: Octenidine treatment — Octenidine dihydrochloride is a cationic surfactant and bis-(dihydropyridinyl)-decane derivative, used in concentrations of 0.1-2.0%. It is similar in its action to the quaternary ammonium compounds, but is of somewhat broader spectrum of activity. Octenidine is currently increasingly used in continental Europe as a substitute for quats or chlorhexidine (with respect to its slow action and concerns about the carcinogenic impurity 4-chloroaniline) in water- or alcohol-based skin, mucosa and wound antiseptics. In aqueous formulations, it is often potentiated with addition of 2-phenoxyethanol.
  Other Names: Octenisept
  Arms: Octenidine treatment

SUMMARY:
Prevalence of diabetic foot ulcers are reported to be 15% in patients who suffer from diabetes and ulcerations are present in 84% of all diabetes-related amputations. Peripheral neuropathy leading to unperceived trauma seems to be the major cause of diabetic foot ulcers with 45-60% of ulcers to be considered merely neuropathic and 45% of mixed, neuropathic and ischemic etiology. Ulceration of lower limb is one of the most common complications related with diabetes and one of the major causes for hospitalization of diabetic patients. The most significant contributors to diabetic lower limb ulceration are neuropathy, deformity, uncontrolled elevated plantar pressure, poor glycemic status, peripheral vascular disease, male gender and duration of diabetes. Treatment of lower limb ulcers imposes an enormous burden on health care resources worldwide, and at least 33% of all expenses are spent to treat diabetic ulcers manifested as a complication of diabetes.

Although at least 170 topical wound care products are available, evidence of the superiority of one over another is tenuous, well-designed randomized, controlled trials are rare, and the number of case-control or observational studies is limited. In recent years, salve prepared from Norway spruce (Picea abies) resin has successfully been used in medical context to treat both acute and chronic wounds and ulcers of various origins. The objective of this prospective, randomized and controlled clinical trial is to investigate healing rate and healing time of neuropathic diabetic foot ulcer in patients, who are suffering from infected fore- or mid-foot ulceration (PEDIS-classification ≥ Grade II; 19) originated from Type I or II diabetes, and in patients whose diabetic ulcerations are candidates for topical treatment with resin (Study treatment) or octenidine (Control treatment). In addition, factors contributing with delayed healing of ulceration, antimicrobial properties, safety and cost-effectiveness of the resin salve treatment and control treatment will be analyzed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES

Primary objectives are:

* to scrutinize complete healing of neuropathic diabetic foot ulceration over time.
* to analyze successful eradication rate of pathogenic bacteria from the ulcers within the study period as documented by negative swab culture.
* to analyze the rate of ulcers with 50% decrease in ulcer size and disappearing of clinical signs of infection over time.

SECONDARY OBJECTIVES

Secondary objectives are:

* to assess potential contributors to delayed ulcer healing.
* to study the safety and compliance related with the treatment methods.
* to estimate the overall costs of the ulcer treatment with the resin salve treatment or octenidine treatment.

INCLUSION AND EXCLUSION CRITERIA

Inclusion criteria are:

* an adult patient (18-80 years) with infected neuropathic foot ulceration due to type I or II diabetes.
* PEDIS-classification ≥ Grade II.

Exclusion criteria are:

* a patient whose life expectancy is less than 6 months.
* an ulceration of ischemic or neuroischemic origin.
* presence of systemic inflammatory response signs.
* heel ulceration.
* presence of osteomyelitis.
* pregnancy.
* known hypersensitivity to any of the ingredient including in the study or control treatment products. - a patient who is unable to give informed consent.
* a patient who has an advanced malignant disease.

METHODS Patient selection Altogether 40 adult patients (18 - 80 years) suffering from infected neuropathic fore- or mid-foot ulceration originated from type I or II diabetes (PEDIS-classification ≥ Grade II) are randomly allocated into two groups (n = 20 patients / group) to receive either topical resin salve treatment or topical octenidine treatment for an appropriate diabetic ulceration. The patients who are recruited to the current study, are selected by the physicians, who are specialized in the treatment of diabetes and its complications. Treatment is commenced and followed-up at the outpatient clinic of the Diabetic Foot Clinic Regional Diabetic Centre, Department of Hypertension and Diabetology, Gdansk, Poland. Informed consent will be obtained from all patients.

FOLLOW-UP Demographics, clinically relevant medical, and follow-up data is gathered on the Clinical Report Form (CRF) by the responsible physicians for every patient at the beginning of the study, and within the every visit at the Diabetic Foot Clinic of the Regional Diabetic Centre until the study ends at six months later, at last. Thus, all recruited patients visit at the Diabetic Foot Clinic: 1. in the beginning of the study, and at 1, 2, 3, and 4 week time-points thereafter. After that, consecutive visit for every 3 to 4 weeks are arranged until the ends after the 6 months from the initiation. If the patient's clinical situation requires more frequent visits at the Diabetic Foot Clinic, those are arranged on the basis of the decision of research physician.

If the ulcer healing takes less than 6 months, the last follow-up information on the CRF is filled when the ulcer is considered being fully healed (primary objective is achieved). If the ulcer is not fully healed in 6 months, the treatment is considered unsuccessful, and follow-up is discontinued (primary objective is not achieved). Photographs are taken within every control visit at the outpatient department. Any notable improvement, deterioration, or any factor that might contribute with the ulcer healing during the follow-up, e.g. mechanical / surgical ulcer revision, cleansing, or antibiotic treatment will be registered on the CRF: Thus, CRF includes the details of:

* size of the ulcer [width (mm) x length (mm) x depth (mm)].
* signs of infection.
* swab culture.
* plain x-ray.
* erythrocyte sedimentation rate (ESR).
* C-reactive protein (CRP).
* full blood count.
* photographs with an appropriate measure.
* use of antibiotics.
* rate of dressing changes.
* potential side-effects (i.e. signs of hypersensitivity or allergic reaction).
* the use of off-loading shoe, and any specific notes or observations during the treatment period.

SAFETY ISSUES Hypersensitivity or allergy for resin or control treatment is taken into account, and if any symptoms of allergic reactions i.e. contact dermatitis appear, the study is discontinued for this particular patient.

ELIGIBILITY:
Inclusion Criteria:

* an adult patient (18-80 years) suffering from infected neuropathic fore- or mid-foot ulceration originated from type I or II diabetes (PEDIS-classification ≥ Grade II).

Exclusion Criteria:

* a patient whose life expectancy is less than 6 months
* an ulceration of ischemic or neuroischemic origin
* presence of systemic inflammatory response signs
* heel ulceration
* presence of osteomyelitis
* pregnancy
* known hypersensitivity to any of the ingredient including in the study or control treatment products
* a patient who is unable to give informed consent
* a patient who has an advanced malignant disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Wound healing | Within 6 months
  To scrutinize complete healing of neuropathic diabetic foot ulceration over time.

SECONDARY OUTCOMES:
Eradication of bacteria | Within six months
  To analyze successful eradication rate of pathogenic bacteria from the ulcers within the study period as documented by negative swab culture.

OTHER OUTCOMES:
Wound healing and infection | Within six months
  To analyze the rate of ulcers with 50% decrease in ulcer size and disappearing of clinical signs of infection over time.

CONTACTS AND LOCATIONS:
Overall Officials: Janne J. Jokinen, MD, PhD, Study Chair — Repolar Pharmaceuticals Oy
Locations (1):
- Diabetic Foot Clinic Regional Diabetic Centre, Department of Hypertension and Diabetology, Gdansk, Gdańsk, Poland

REFERENCES:
- [Background] Reiber GE, Vileikyte L, Boyko EJ, del Aguila M, Smith DG, Lavery LA, Boulton AJ. Causal pathways for incident lower-extremity ulcers in patients with diabetes from two settings. Diabetes Care. 1999 Jan;22(1):157-62. doi: 10.2337/diacare.22.1.157. PMID 10333919
- [Background] Frykberg RG. Diabetic foot ulcers: pathogenesis and management. Am Fam Physician. 2002 Nov 1;66(9):1655-62. PMID 12449264
- [Background] Akbari CM, Macsata R, Smith BM, Sidawy AN. Overview of the diabetic foot. Semin Vasc Surg. 2003 Mar;16(1):3-11. doi: 10.1053/svas.2003.50001. No abstract available. PMID 12644970
- [Background] Frykberg RG, Zgonis T, Armstrong DG, Driver VR, Giurini JM, Kravitz SR, Landsman AS, Lavery LA, Moore JC, Schuberth JM, Wukich DK, Andersen C, Vanore JV; American College of Foot and Ankle Surgeons. Diabetic foot disorders. A clinical practice guideline (2006 revision). J Foot Ankle Surg. 2006 Sep-Oct;45(5 Suppl):S1-66. doi: 10.1016/S1067-2516(07)60001-5. PMID 17280936
- [Background] Driver VR, Fabbi M, Lavery LA, Gibbons G. The costs of diabetic foot: the economic case for the limb salvage team. J Vasc Surg. 2010 Sep;52(3 Suppl):17S-22S. doi: 10.1016/j.jvs.2010.06.003. PMID 20804928
- [Background] Sipponen A, Jokinen JJ, Lohi J. Resin salve from the Norwegian spruce tree: a 'novel' method for the treatment of chronic wounds. J Wound Care. 2007 Feb;16(2):72-4. doi: 10.12968/jowc.2007.16.2.26999. No abstract available. PMID 17319621
- [Background] Sipponen A, Jokinen JJ, Sipponen P, Papp A, Sarna S, Lohi J. Beneficial effect of resin salve in treatment of severe pressure ulcers: a prospective, randomized and controlled multicentre trial. Br J Dermatol. 2008 May;158(5):1055-62. doi: 10.1111/j.1365-2133.2008.08461.x. Epub 2008 Feb 16. PMID 18284391
- [Background] Rautio M, Sipponen A, Peltola R, Lohi J, Jokinen JJ, Papp A, Carlson P, Sipponen P. Antibacterial effects of home-made resin salve from Norway spruce (Picea abies). APMIS. 2007 Apr;115(4):335-40. doi: 10.1111/j.1600-0463.2007.apm_548.x. PMID 17504300
- [Background] Rautio M, Sipponen A, Lohi J, Lounatmaa K, Koukila-Kahkola P, Laitinen K. In vitro fungistatic effects of natural coniferous resin from Norway spruce (Picea abies). Eur J Clin Microbiol Infect Dis. 2012 Aug;31(8):1783-9. doi: 10.1007/s10096-011-1502-9. Epub 2011 Dec 17. PMID 22179415
- [Background] Sipponen A, Laitinen K. Antimicrobial properties of natural coniferous rosin in the European Pharmacopoeia challenge test. APMIS. 2011 Oct;119(10):720-4. doi: 10.1111/j.1600-0463.2011.02791.x. Epub 2011 Jul 18. PMID 21917009
- [Background] Sipponen A, Peltola R, Jokinen JJ, Laitinen K, Lohi J, Rautio M, Mannisto M, Sipponen P, Lounatmaa K. Effects of Norway spruce (Picea abies) resin on cell wall and cell membrane of Staphylococcus aureus. Ultrastruct Pathol. 2009;33(3):128-35. doi: 10.1080/01913120902889138. PMID 19479653
- [Background] Lipsky BA, Berendt AR, Cornia PB, Pile JC, Peters EJ, Armstrong DG, Deery HG, Embil JM, Joseph WS, Karchmer AW, Pinzur MS, Senneville E. 2012 infectious diseases society of america clinical practice guideline for the diagnosis and treatment of diabetic foot infections. J Am Podiatr Med Assoc. 2013 Jan-Feb;103(1):2-7. doi: 10.7547/1030002. PMID 23328846
- [Background] Brolmann FE, Ubbink DT, Nelson EA, Munte K, van der Horst CM, Vermeulen H. Evidence-based decisions for local and systemic wound care. Br J Surg. 2012 Sep;99(9):1172-83. doi: 10.1002/bjs.8810. Epub 2012 Jul 6. PMID 22777856
- [Background] Hubner NO, Siebert J, Kramer A. Octenidine dihydrochloride, a modern antiseptic for skin, mucous membranes and wounds. Skin Pharmacol Physiol. 2010;23(5):244-58. doi: 10.1159/000314699. Epub 2010 May 18. PMID 20484966
- [Background] Krishna BV, Gibb AP. Use of octenidine dihydrochloride in meticillin-resistant Staphylococcus aureus decolonisation regimens: a literature review. J Hosp Infect. 2010 Mar;74(3):199-203. doi: 10.1016/j.jhin.2009.08.022. Epub 2010 Jan 8. PMID 20060619
- [Background] Moher D, Schulz KF, Altman DG. The CONSORT statement: revised recommendations for improving the quality of reports of parallel-group randomised trials. Lancet. 2001 Apr 14;357(9263):1191-4. PMID 11323066